CLINICAL TRIAL: NCT01542320
Title: Application of Therapeutic Microbiology to Improve Immunogenicity
Brief Title: Effect of Probiotic Supplementation on Immune Function in Healthy Infants
Acronym: ProBoost
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Principal Investigator, Andi L. Shane, MD, Assistant Professor of Pediatrics, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: IRB00055040; ProBoost (Other: Other)
Record Dates: First submitted 2012-02-21; First posted 2012-03-02 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2014-11

CONDITIONS: Inflammation
Keywords: probiotic; Lactobacillus reuteri DSM 17938; healthy infants
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic (Experimental): Lactobacillus reuteri DSM 17938
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM 17938
- Placebo (Placebo Comparator): Solution without the active probiotic Lactobacillus reuteri
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri DSM 17938 — 1 x 10e8 colony forming units in 5 drops (0.17ml)daily from study enrollment to study conclusion. Duration based on rotavirus vaccine administration.
  Other Names: BioGaia infant drops
  Arms: Probiotic
Other: Placebo — Solution without active Lactobacillus reuteri
  Other Names: Inactive solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to understand how a probiotic might change the immune response of healthy infants.

DETAILED DESCRIPTION:
PROBLEM OF INTEREST: Lactic acid bacteria known as probiotics have been given to children and adults to prevent and treat gastrointestinal infections and to maintain intestinal health. This pilot study will collect information (biomarkers) of inflammation and immune response from healthy infants.

HOW THE PROBLEM WILL BE STUDIED: The investigators will give an active Lactobacillus-containing probiotic or an inactive placebo without Lactobacillus to 38 healthy infants in the metropolitan Atlanta area from 2 weeks before until 2 weeks after they complete their rotavirus vaccine series. Half will be assigned to receive the active probiotic, half to receive the placebo. Neither the investigators nor the parent/ guardian of the study subject will know whether their infant is receiving the probiotic or placebo. A teaspoon of blood and a stool sample will be collected from each infant before they start taking the active probiotic or placebo and 2 weeks after they complete their rotavirus vaccine series. Each infant will receive the probiotic or placebo product for 2 weeks before starting their rotavirus vaccine series until 2 weeks after they complete their rotavirus vaccine series. The blood and stool samples will be examined for levels of inflammatory markers and measures of immune response. The stool samples may be stored for the later study of probiotic bacteria as well as for other bacteria and viruses. These results will help to determine if this Lactobacillus containing probiotic has an effect on immune response and inflammation in healthy infants.

HOW RESEARCH WILL ADVANCE SCIENTIFIC KNOWLEDGE AND HUMAN HEALTH: This study will provide new information about the impact of giving a Lactobacillus-containing probiotic supplement to healthy infants. CURRENT STANDARD OF CARE: The current standard of care is for infants to receive a probiotic at the discretion of their caregiver. By studying probiotic administration in a controlled way with a fixed dose schedule and a well categorized probiotic, and measuring blood and stool markers, the investigators hope to better understand the impact of a probiotic on immune response and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infant
* Eligible for rotavirus immunization series
* No recognized immunodeficiency
* Ability to comply with study procedures

Exclusion Criteria:

* Ineligible for rotavirus immunization series
* Recognized immunodeficiency
* Inability to comply with study procedures

Ages: 6 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Biomarkers of immune response | Between 18 and 32 weeks of age

CONTACTS AND LOCATIONS:
Overall Officials: Andi L Shane, MD, MPH, MSc, Principal Investigator — Emory University
Locations (1):
- Emory Children's Center, Atlanta, Georgia, United States